CLINICAL TRIAL: NCT01158027
Title: Evaluating Walking Kinetic of Children Who Suffer Central Nervous System (CNS)
Brief Title: Evaluating Walking Kinetic of Children Who Suffer Central Nervous System (CNS) Damage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofer Keren, MD, Sheba Medical Center
Other Study IDs: SHEBA-10-7999-OK-CTIL
Record Dates: First submitted 2010-07-04; First posted 2010-07-08 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Walking Performance

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children
  Interventions: Other: gait evaluation

INTERVENTIONS:
Other: gait evaluation — The children will asked to walk under different conditions: (1) walking at a self-selected speed faster and slower on the GAITRite® system and on a treadmill and while listening and to a metronomeQuoting.

SUMMARY:
The goal of the present study is to look at the effect of changing walking parameters on the dynamic walking characteristics among children post severe traumatic brain injury, and typically developed controls.

ELIGIBILITY:
Inclusion Criteria:

1. post-severe closed head injury (Glasgow Coma Scale [GCS] score at admission to emergency room of ≤8) [Kathryn 2008].
2. at least one year post trauma.
3. ages 7 to 13 years.
4. independent ambulation (foot orthoses permitted).

Exclusion Criteria:

1. had received botulinum toxin for spasticity management or had undergone orthopedic surgery in the past six months.
2. unable to follow simple instructions.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fifteen children post-TBI and fifteen typically control.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-10